CLINICAL TRIAL: NCT06646380
Title: The Importance of the Interplay Between Physical Fitness, Sleep Quality, Dynamic Balance and Exercise Intervention in Aged People
Brief Title: Physical Fitness, Sleep Quality, Dynamic Balance and Exercise in Aged People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Politécnico de Bragança (Other)
Collaborators: Research Center for Active Living and Wellbeing (Unknown); University of Alcala (Other)
Responsible Party: Principal Investigator, Pedro Miguel Gomes Forte, Professor, University of Alcala
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 501020
Record Dates: First submitted 2024-10-09; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Aged 60 Years or Older; Aged Healthy Volunteer
Keywords: aged; physical fitness; body composition; sleep quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multicomponent Training (Experimental): Participants will be instructed to maintain normal daily life activities to prevent physical inactivity. Inclusion criteria will involve individuals over 65 years old, independent in daily activities, and without chronic diseases requiring pharmacological treatment affecting the experimental protocol, while exclusion criteria included failure to attend more than 25% of training sessions, failure to attend more than four consecutive sessions, or missing evaluation sessions. Participants will be randomly assigned to either the experimental group (EG ≈ 30) or control group (CG ≈ 30). Experimental group will be followed-up during the exercise sessions.
  Interventions: Behavioral: Multicomponent Training
- Control Group (Placebo Comparator): The CG were instructed to maintain their daily life routines. However, the typical profile of this group was that the participants were regularly physically active people. Most participate in municipal activities like nature walking, physical activity sessions including dance (casually), board and card games, and traditional games (Bocce, Adapted Bowling, and darts).
  Interventions: Other: Maintenance

INTERVENTIONS:
Behavioral: Multicomponent Training — The multicomponent training (MCT) program comprised aerobic, resistance, flexibility, and balance exercises, following recommendations by Carvalho et al. (23). Sessions lasted 50 to 60 minutes, including warm-up, aerobic exercise, resistance training, balance training, and cool-down. Training intensity gradually increased over time. The experimental group will have three 60-minute sessions weekly for 32 weeks, while the control group will not participate in any exercise program, but they will maintain the daily physical activity. Both groups will be evaluated at two time points: initial assessment (M1) at the start of training and final assessment (M2) after 32 weeks
  Arms: Multicomponent Training
Other: Maintenance — Participants were instructed to maintain daily life activities regarding physical activity.
  Arms: Control Group

SUMMARY:
Nowadays, the sedentary lifestyles and aging related problem to well-being, have a significant impact on of physical fitness, quality of life, and sleep in elderlies. The regular exercise is of higher importance crucial for maintaining overall health and delay some ageing-related declines in physical fitness. The multicomponent training (MCT) programs, include exercises to promote endurance, strength, flexibility, and balance. The MCT are typically effective to improve physical fitness, quality of life, sleep, and balance in older populations. Notably, in visually impaired older adults, lower limb function is closely linked to fall risk. Improving the muscular strength and bone health enhances the balance and the gait. Additionally, it is possible to find associations between sleep quality, frailty, and quality of life among older adults, highlighting the interplay between sleep, physical health, and overall well-being in aging populations. Another study, highlighted that the socioeconomic status and sleep quality's influence on the prevalence of multimorbidity in older adults, underscoring the broader health implications of sleep disturbances in aging populations.

The principal objective of the current PhD research project is to assess the effects of a multicomponent training programs on critical variables such as physical fitness, sleep quality, and dynamic balance in older adults.

DETAILED DESCRIPTION:
To successfully close this research project and in agreement with the stablished objectives and hypothesis, a compendium of three future published articles as part of the thesis. The first article will be a review about the relationships between exercise, sleep quality, physical fitness and dynamic balance. This review article will answer the first hypothesis and objective. The second article, will be an observational research article. The data from the baseline evaluation will allow to run artificial intelligence algorithms, intending to predict the dynamic balance variance based on physical fitness and quality of sleep. This article aims to identify the variables that mostly explain the dynamic balance based on body composition and antropometrics, sleep quality and physical fitness. This article will answer to the second hypothesis and objective. The third article will be a randomized controlled trial article. This part of the research will seek to understand the effects of (8 months) multicomponent exercise training program in antropometric and body composition, sleep quality, physical fitness effects and dynamic balance.

Study design: The present project will adopt a longitudinal approach wherein volunteers will be briefed about the study objectives and protocol and were required to provide informed consent, adhering to the Helsinki Declaration guidelines. Participants were instructed to maintain normal daily life activities to prevent physical inactivity. Inclusion criteria will involve individuals over 65 years old, independent in daily activities, and without chronic diseases requiring pharmacological treatment affecting the experimental protocol, while exclusion criteria included failure to attend more than 25% of training sessions, failure to attend more than four consecutive sessions, or missing evaluation sessions. Participants will be randomly assigned to either the experimental group (EG ≈ 30) or control group (CG ≈ 30). The multicomponent training (MCT) program comprised aerobic, resistance, flexibility, and balance exercises. Sessions lasted 50 to 60 minutes, including warm-up, aerobic exercise, resistance training, balance training, and cool-down. Training intensity gradually increased over time. The experimental group will have three 60-minute sessions weekly for 32 weeks, while the control group will not participate in any exercise program, but they will maintain the daily physical activity. Both groups will be evaluated at two time points: initial assessment (M1) at the start of training and final assessment (M2) after 32 weeks. The Physical fitness will be assessed using the Rikli and Jones Senior Fitness Test. The Sleep quality evaluated by the Pittsburgh Sleep Quality Index (PSQI). Dynamic balance will be assessed using the Timed Up and Go Test (TUG). Additionally, body composition before and after the training program will be evaluated by bioimpedance.

Physical Fitness: The Rikli and Jones Senior Fitness Test will be used to assess the physical fitness. The following tests will be used: limb strength and endurance of lower (30-s chair stand and seat, by the number of repetitions) and upper limbs (arm curl with 2 kg dumbbell); lower flexibility (chair sit-and-reach, in centimeters) and superior flexibility (back scratch, in centimeters); physical mobility, speed, agility and dynamic balance (stand up the chair and run 8-ft up-and-go returning and seat on the chair, measured in seconds); and aerobic endurance (2 min step test, rising and counting the repetitions, when the knee reaches the hip level).

Sleep Quality: The Pittsburgh Sleep Quality Index (PSQI) will be used to assess the sleep quality. This instrument consists in a set of 19 self-reported questions is divided into seven subcategories, covering various aspects of sleep experience such as perceived sleep quality, time taken to fall asleep, duration of sleep, efficiency of sleep, disturbances during sleep, use of sleep aids, and daytime functionality.

Additionally, five extra questions, assessed by the respondent's roommate or bed partner, are included for clinical assessment but do not contribute to the scoring process. The instrument's psychometric properties using a sample of individuals ranging in age from 24 to 83 years. There are some literature that examined the psychometric characteristics of the scale, the developers' initial assessment revealed an internal reliability of α = .83, a test-retest reliability of .85 for the overall scale, with a sensitivity of 89.6% and a specificity of 86.5%.

Dynamic Balance: The Timed Up and Go Test (TUG) will be used to assess the dynamic balance. The individuals will start in a seated position in a chair with armrests. Upon receiving a verbal cue, they stand up, walk approximately 3 meters (10 feet) at their usual pace, turn around, walk back to the chair, and sit down again. This test evaluates dynamic balance by measuring the time taken (in seconds) to complete the task, reflecting the individual's ability to transition between sitting and standing, walk safely, turn, and return to a seated position, which is indicative of their dynamic balance and mobility. Interpretation of the results is based on the completion time, where shorter times suggest better dynamic balance and mobility, while longer times may indicate limitations in balance and mobility. Typically, measured in seconds, cutoff values for the TUG test may vary depending on factors such as age and health status, but shorter completion times generally signify better dynamic balance and mobility, with completion times of approximately 10 seconds or less considered indicative of good functional mobility and balance in older adults.

ELIGIBILITY:
Inclusion Criteria:

* being aged 60 years or older;
* maintaining functional independence in daily tasks;
* having no severe chronic diseases or medications to sleep that could affect the results:
* do not have significant cardiovascular, muscular, metabolic, or joint complications.

Exclusion Criteria:

* Less than 60 years old.
* Be dependent of caregiver in daily life activities.
* Use medication to sleep or tranquilizers.
* Have cardiovascular, muscular, metabolic or joint diseases.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Sleep Quality | At baseline (0 weeks) and at 32 weeks
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI), a 19-item questionnaire developed by and validated for the Portuguese population. The PSQI items are divided into the following components: 1) subjective sleep quality, 2) sleep latency, 3) sleep duration, 4) habitual sleep efficiency, 5) sleep disturbances, 6) use of sleeping medication, and 7) daytime dysfunction. Each item is scored from 0 to 3, with the total score ranging from 0 to 21; higher scores indicate more severe sleep disturbances. A global score of 5 or higher in two components signifies significant sleep difficulties, while a score in three or more components indicates moderate sleep issues. A total score below 5 indicates good sleep quality, whereas a score above 5 indicates poor sleep quality.

SECONDARY OUTCOMES:
Handgrip strength | At baseline (0 weeks) and at 32 weeks
  Handgrip strength was assessed using a digital with the maximum kilograms-force (kgf)
2-Minute Step Test | At baseline (0 weeks) and at 32 weeks
  The 2-Minute Step Test, where the evaluator set a knee height marker using a measuring tape to measure from the kneecap to the iliac crest, and participants aimed to take as many steps as possible in two minutes, with performance checks at 60 and 90 seconds.
The Seat-to-Stand Test | At baseline (0 weeks) and at 32 weeks
  The The Seat-to-Stand Test required participants to repeatedly sit and stand from a 43 cm highchair for 30 seconds, recording the number of repetitions.
Arm Curl Test | At baseline (0 weeks) and at 32 weeks
  The Arm Curl Test, using a 2 kg dumbbell to perform elbow curls for 30 seconds.
Time-Up-and-Go Test | At baseline (0 weeks) and at 32 weeks
  The Time-Up-and-Go Test involved starting from a seated position on a 43 cm chair, walking quickly around a cone placed 2.44 meters away.
Sit and Reach Test | At baseline (0 weeks) and at 32 weeks
  The Sit and Reach Test, conducted while seated on a 43 cm chair with one leg extended and toes reached
Back Scratch Test | At baseline (0 weeks) and at 32 weeks
  The Back Scratch Test, where participants attempted to touch one hand with the other behind their back (cm)
Five-time sit-to-stand | At baseline (0 weeks) and at 32 weeks
  The five-time sit-to-stand test (sg)
Body Mass | At baseline (0 weeks) and at 32 weeks
  Body Mass (Kg)
Wist circumference | At baseline (0 weeks) and at 32 weeks
  Waist circumference (cm) perimeter.
Hip circumference | At baseline (0 weeks) and at 32 weeks
  Hip circumference (cm) perimeter
Total Fat | At baseline (0 weeks) and at 32 weeks
  Total Fat in Kg and Percentage (%).
Body Water | At baseline (0 weeks) and at 32 weeks
  Body Water (%)
Visceral Fa (a.u.) | At baseline (0 weeks) and at 32 weeks
  Visceral Fat (a.u.) in levels.
Basal Metabolic Rate | At baseline (0 weeks) and at 32 weeks
  Basal Metabolism (Kcal)
Body Mass Index (BMI) | At baseline (0 weeks) and at 32 weeks
  weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Miguel Forte, PhD, Principal Investigator — University of Alcala
Locations (1):
- Instituto Politécnico de Bragança, Bragança, Braganza District, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Solis-Navarro L, Masot O, Torres-Castro R, Otto-Yanez M, Fernandez-Jane C, Sola-Madurell M, Coda A, Cyrus-Barker E, Sitja-Rabert M, Perez LM. Effects on Sleep Quality of Physical Exercise Programs in Older Adults: A Systematic Review and Meta-Analysis. Clocks Sleep. 2023 Mar 23;5(2):152-166. doi: 10.3390/clockssleep5020014. PMID 37092426
- [Background] Rodrigues F, Jacinto M, Figueiredo N, Monteiro AM, Forte P. Effects of a 24-Week Low-Cost Multicomponent Exercise Program on Health-Related Functional Fitness in the Community-Dwelling Aged and Older Adults. Medicina (Kaunas). 2023 Feb 15;59(2):371. doi: 10.3390/medicina59020371. PMID 36837572